CLINICAL TRIAL: NCT05020587
Title: Consulting After Combat: Interviewing Service Members and Veterans to Develop a Therapy to Restore Functioning and Reintegration After Moral Injury Events
Brief Title: Consulting After Combat: Interviewing Veterans to Develop a Therapy to Restore Functioning and Reintegration After Moral Injury Events
Acronym: CAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3495-W; RX003495 (Registry Identifier: eRA Commons)
Record Dates: First submitted 2021-07-12; First posted 2021-08-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Moral Injury; Functional Impairment
Keywords: Moral Injury; Group Psychotherapy; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Two open pilot trials of a novel time-limited potentially morally injurious event (PMIE)-focused therapy group (N ~= 12), led by two therapists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Pilot Trial (Other): Open pilot trial of a group therapy manual.
  Interventions: Behavioral: Open pilot trial of a group therapy manual.

INTERVENTIONS:
Behavioral: Open pilot trial of a group therapy manual. — Open pilot trial of a group therapy manual.

SUMMARY:
Despite the VA's best efforts to treat the psychosocial impact of war, many combat Veterans report lingering difficulty reintegrating into meaningful post-deployment lives. War is among the most extreme forms of human experience but, for many, wartime trauma was treated using models transported from civilian single-incident trauma contexts. Veterans have unique needs and experiences that require culturally responsive and sensitive conceptualizations and treatments. Patient-centered care is improved by providing multiple effective treatment options and this project, if successful, could have a significant impact on VA care. This CDA-2 project has the potential to offer innovative treatment for traumatized combat Veterans who otherwise may not find full relief from PTSD. Clinical research practice will be advanced by employing state-of-the-art user-centered design methods combined with expert clinical feedback to develop an effective and usable group treatment manual that will meet VA needs.

DETAILED DESCRIPTION:
Approximately 25% of combat Veterans with Posttraumatic Stress Disorder (PTSD) seek treatment for traumas that involve potentially morally injurious events (PMIE) rather than danger-based traumas. PMIEs are more strongly associated with functional and psychiatric impairment than life-threat-based combat. Veterans report that PMIEs disrupt their sense of identity and meaning, ability to connect with and trust others, and engender disturbing guilt, shame, rage, and disgust. The sequelae of exposure to PMIEs, otherwise known as moral injury, may explain variance in post-deployment recovery and is a potential unaddressed treatment target. Existing first-line treatments may be limited because they were derived from civilian contexts, poorly fit the war zone context, and do not allow Veterans to discuss the details of the PMIEs with other Veterans. This project will develop a relational dynamic-based group therapy treatment manual that will target functioning and quality of life among Veterans who are impacted by high magnitude PMIEs. The goal of this relational dynamic trauma therapy is to help Veterans identify connections between their current symptoms and their experiences in combat/PMIEs, their current life stressors and relationships, and the historical factors that carry person-specific meaning to their trauma/PMIE. These explorations take place in the presence of attuned and sympathetic others who can resonate to the experience and the affect being expressed. Symptom reduction occurs through increasing the Veteran's capacity to consciously reflect on their experiences and develop an integrated self-awareness of the various factors that affect their mental states. The result is greater self-reflection, less avoidance, and greater adaptive incorporation of life experiences and their aftermath and meanings into one's inner world. This CDA-2 will employ innovative user-centered design methods that continuously gather user experiences during treatment development, with the goal of increased effectiveness and usability. User feedback will be synthesized with formative feedback from a clinical expert panel. This objective will be accomplished by pursuing these specific aims: Aim 1: Discover user needs and preferences as well as treatment-engagement barriers and facilitators from the perspectives of PMIE-impacted Veterans and VA trauma clinicians. Aim 2: Design a treatment manual and refine it using feedback from Veterans, trauma clinicians, and an expert clinical advisory board. Aim 3: Conduct two rapid prototyping open trials (i.e., tangibly testing treatment approaches using a prototype manual) with PMIE-impacted Veterans (N = ~12), and iteratively revise the manual based on Veteran, provider, and clinical expert panel feedback, with the following hypothesis: The treatment manual will meet usability, feasibility, learnability, and acceptability criteria.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit 12 potentially morally injurious event (PMIE)-impaired Veterans.
* Potential participants include:

  * male and female
  * English-speaking Veterans
  * 18 years of age or older
  * enrolled in Central Texas Veterans Healthcare System
  * with a service record of combat deployments
* Participants must:

  * comprehend and sign the informed consent form
  * if they report a PMIE as their worst trauma
  * 3 on the MIOS functional impairment item
  * if they score 10 on the SDS

Exclusion Criteria:

* Veterans will be excluded from the study if they have either:

  * untreated substance abuse disorder
  * severe suicidal or homicidal ideation, defined using the C-SSRS
  * <18 on the MOCA, indicating potential for more than mild cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | One-month following the conclusion of the pilot trial and 6-months following the conclusion of the pilot trial.
  The AIM will be descriptively analyzed, and the mean and standard deviation; mean scores >/ 4 will indicate acceptability.
Implementation Appropriateness Measure (IAM) | One-month following the conclusion of the pilot trial and 6-months following the conclusion of the pilot trial.
  The IAM is a 4-item measure. The IAM will be descriptively analyzed, and the mean and standard deviation will be reported; mean scores >/ 4 will indicate appropriateness (via the IAM).
Feasibility of Intervention Measure (FIM) | One-month following the conclusion of the pilot trial and 6-months following the conclusion of the pilot trial.
  The FIM is a 4-item measure. The FIM will be descriptively analyzed, and the mean and standard deviation will be reported; mean scores >/ 4 will indicate feasibility (via the FIM).

SECONDARY OUTCOMES:
Moral Injury Outcome Scale (MIOS) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  The 14-item MIOS assesses exposure to a PMIE, prior month multidimensional outcomes associated with the PMIE, and prior month PMIE-related functional impairment. Items are rated on a Likert-style scale ranging from 0 (strongly disagree) to 4 (strongly agree). Higher scores are indicative of more moral injury. Change in moral injury from pre- to post-intervention will be examined.
Change in Posttraumatic Stress Disorder Checklist-5 (PCL-5) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  PTSD will be measured with the widely used 20-item Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5), which assesses severity of each DSM-5 PTSD symptom using a Likert-style ranging from 0 (not at all) to 4 (extremely). A total score of 31-33 is suggestive of a PTSD diagnosis. Change in PTSD symptom severity from pre- to post-intervention will be examined.
Change in Beck Depression Inventory-II (BDI-II) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  Depression will be measured with the 21-item Beck Depression Inventory-II (BDI-II), which uses a Likert-style scale ranging from 0 to 3. Lower scores are indicative of less severe depression. Change in depressive symptoms from pre- to post-intervention will be examined.
Change in Beck Scale for Suicide Ideation (BSS) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  Suicidal ideation will be measured using the Beck Scale for Suicide Ideation (BSS), which is extensively used in treatment studies of suicidal individuals. The BSS is rated on a Likert-style scale ranging from 0 to 3, which lower scores indicative of less severe suicidal ideation. Change in suicidal ideation from pre- to post-intervention will be examined.
Change in Religious and Spiritual Struggles Scale (RSSS) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  The 26-item RSSS assesses six domains including moral and doubt struggles using a Likert-style scale ranging from 0 to 5.
Change in Moral Injury Events Scale (MIES) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  The MIES is a 9-item measure that assess perceptions of potentially morally injurious events. Items are rated on a 1 (Strongly agree) to 6 (strongly disagree) Likert-style scale, and lower scores are indicative of more moral injury. Change in endorsement of moral injury events will be assessed from pre- to post-intervention.
Group Cohesion Scale-Revised (GCS) | Post intervention (approximately 6 weeks)
  The 25-item Group Cohesion Scale-Revised measures group functioning on a Likert-style ranging from 0 (low) to 4 (strongly agree). Higher scores are indicative of greater group cohesion.
Change in Brief Expressions of Moral Injury Scale (EMIS) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  The Brief EMIS is a 6-item scale that assesses moral injury event-related guilt, shame, and related outcomes. Items are rated on a Likert-style on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher scores indicate greater moral injury. Change in moral injury will be assessed from pre- to post-intervention.
Brief Inventory of Psychosocial Functioning (bIPF) | Pre intervention (Baseline), post intervention (approximately 6 weeks), and following the conclusion of the intervention, up to 6 months
  The bIPF is a 6-item measures that assesses six domains of psychosocial functioning (i.e., romantic relationships, relationships with children, relationships with family, work, activities of daily living, training/education) on a 7-point Likert-style 0 (not at all) - 6 (extremely) scale. Domains that are not applicable are indicated as NA.

OTHER OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | Eligibility screening (pre-intervention)
  The C-SSRS is the VA-mandated suicide screening tool used in primary care and mental health clinics across the VA. The C-SSRS assesses lifetime and past-month suicidal ideation, intent, plans, and behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Beth Frankfurt O'Brien, PhD, Principal Investigator — Central Texas Veterans Health Care System, Temple, TX
Locations (1):
- Central Texas Veterans Health Care System, Temple, TX, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT05020587/ICF_000.pdf